CLINICAL TRIAL: NCT00002858
Title: PHASE III STUDY COMPARING TWO DOSES OF INDUCTION CHEMOTHERAPY FOLLOWED BY ALTERNATION OF CHEMOTHERAPY AND RADIOTHERAPY IN LIMITED SMALL CELL LUNG CANCER
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065122; FRE-CPC014; EU-96009
Record Dates: First submitted 1999-11-01; First posted 2004-03-12 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-05

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Cyclophosphamide; Doxorubicin; Etoposide; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells. It is not yet known which treatment regimen is more effective for small cell lung cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of combination chemotherapy using two different doses of cyclophosphamide followed by alternating chemotherapy and radiation therapy in treating patients with small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effect on 2-year disease-free survival of two different doses of cyclophosphamide as part of first induction chemotherapy followed by alternating chemotherapy and chest irradiation in patients with limited stage small cell lung cancer.

OUTLINE: This is a randomized study. Patients are stratified by participating institution. All patients receive 2 courses of induction chemotherapy with doxorubicin, etoposide, cisplatin, and cyclophosphamide. For the first course, one group of patients receives a lower dose of cyclophosphamide than the other group. Both groups receive the same, and still lower, dose of cyclophosphamide during the second course. Beginning 1 week after the completion of induction therapy, patients receive 3 alternating courses each of radiotherapy to the mediastinal and supraclavicular areas delivered over 10-12 days and chemotherapy as in the second course of induction. Each course is initiated after a 1-week rest. Patients receive a final chemotherapy course beginning 4 weeks after the previous chemotherapy course. Patients are followed every 6 months for survival.

PROJECTED ACCRUAL: A total of 280 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven small cell lung cancer with no distant metastases Size of initial lesion suitable for total irradiation Positive subclavicular nodes allowed No malignant pleural effusion No extension into contralateral lung

PATIENT CHARACTERISTICS: Age: Under 70 Performance status: Karnofsky 60%-100% Hematopoietic: WBC greater than 2,000 Platelets greater than 125,000 Hepatic: Not specified Renal: Creatinine less than 1.1 mg/dL (100 micromoles/L) Cardiovascular: No myocardial infarction within 6 months No other cardiovascular disease that precludes protocol treatment Other: No hearing loss No prior or concurrent malignancy except: Basal cell skin carcinoma In situ carcinoma of the cervix Accessible for follow-up

PRIOR CONCURRENT THERAPY: No prior chemotherapy, radiotherapy, or surgery

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 1993-03

CONTACTS AND LOCATIONS:
Overall Officials: Thierry L. Le Chevalier, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (19):
- France (19):
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - Centre Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Hopital Antoine Beclere, Clamart
  - Centre Hospitalier Sud Francilien - Site Corbeil, Corbeil
  - Hopital Intercommunal De Creteil, Créteil
  - Hopital De La Trouhade, Dijon
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - C.H. General Andre Boulloche, Montbéliard
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - Hopital Haut Leveque, Pessac
  - C.H. De Saumur, Saumur
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - CHRU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif